CLINICAL TRIAL: NCT01188525
Title: Pharmacokinetic of Ten Parent Drugs and Their Metabolits in Order to Characterise Individual Metabolic Profile
Brief Title: Pharmacokinetic Study to Characterize Individual Metabolic Profile
Acronym: CIME1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: Nuclear Energy Commission (CEA) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C09-04; 2009-014866-24 (EudraCT Number)
Record Dates: First submitted 2010-07-09; First posted 2010-08-25 (Estimated); Last update posted 2025-09-03 (Actual); Status verified 2012-05

CONDITIONS: Healthy Volunteers
Keywords: pharmacokinetics; enzymes; metabolism prediction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: 10 parents drugs adminstration — A single and concomittant administration of 10 parent drugs will be performed: Acetaminophene, cafeine, dextrometorphan, digoxin, memantine,midazolam, omeprazole, repaglinide, rosuvastatine, tolbutamide.

SUMMARY:
The study aims to descibe the pharmacokinetics of 10 substrates of enzymes involved in drug metabolism and their metabolites, after administration singly and simultaenously at predefined doses in 10 health volunteers.

DETAILED DESCRIPTION:
The aim of this study is to test the administration of combination of substrates and thereby to characterise simultaneously the main enzymes and transporters involved in drug metabolism. The doses of substrates administered will first assessed in terms of safety and their appropriateness for determination of pharmacokinetic parameters. Ten volunteers will be used, this number having been defined in view of the aims of this proof-of-concept pilot study,ie,safety and determination of pharmacokinetic parameters. The number was not the result of statistical calculation.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers

Exclusion Criteria:

* pregnancy

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2010-08; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters | one week
  The aim endpoint is based on the main pharmacokinetic parameters of each subject for all substrates and all metabolites. These main parameters are the area under the curve (AUC), the maximum concentration (Cmax), the half-life (T1/2)and the ratios of AUCs of the substrate and metabolites

SECONDARY OUTCOMES:
Tolerance of the concomittant administration of the 10 drugs: 1/number of volunteers with grade 4 adverse events 2/ number of volunteers with any adverse event, (grade 1 to grade 4) | one week
  All clinical and biological adverse events will be recorded within the 7 days following drug administration.
pharmacokinetic | one week
  To determine which sampling times will provid the most pharmacokinetic information on the most compounds
Genotypes | one month
  Depending on the genotypes of the volunteers included, to evaluate the influence of these genotypes ont he pharmacokinetics of the substrates and their metabolites

CONTACTS AND LOCATIONS:
Overall Officials: DUVAL Xavier, doctor, Principal Investigator — Center of clinical investigation
Locations (1):
- Center of clinical investigation, Paris, France

REFERENCES:
- [Background] Lenuzza N, Duval X, Nicolas G, Thevenot E, Job S, Videau O, Narjoz C, Loriot MA, Beaune P, Becquemont L, Mentre F, Funck-Brentano C, Alavoine L, Arnaud P, Delaforge M, Benech H. Safety and pharmacokinetics of the CIME combination of drugs and their metabolites after a single oral dosing in healthy volunteers. Eur J Drug Metab Pharmacokinet. 2016 Apr;41(2):125-38. doi: 10.1007/s13318-014-0239-0. Epub 2014 Dec 3. PMID 25465228